CLINICAL TRIAL: NCT05772481
Title: Interest of PET-MRI in the Evaluation of the Response After Neoadjuvant Treatment of Locally Advanced Rectal Adenocarcinoma
Acronym: TEPIREC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-007
Record Dates: First submitted 2023-02-08; First posted 2023-03-16 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult population with rectal cancer
  Interventions: Other: PET-MRI

INTERVENTIONS:
Other: PET-MRI — Each patient will have a pre-treatment PET-MRI (PET-MRI 1) within 21 days before the start of treatment.
  Induction chemotherapy may be performed at another center than the investigating center.
  After 3 cycles of induction chemotherapy and before the 4th cycle, a second PET MRI (PET MRI 2) will be performed. In patients who have received less than 3 cycles of induction chemotherapy, this mid-therapy PET-MRI will not be performed.
  A 3rd PET-MRI will be performed prior to radiation therapy (PET-MRI 3). A final MRI PET (MRI PET 4) will take place before surgery.
  A total of 4 PET MRI scans will be performed.

SUMMARY:
With 50 patients included, this trial would be the largest pilot study evaluating the value of MRI PET in locally advanced rectal cancer. On the other hand, it would be the only pilot study performing several MRI PET during neoadjuvant treatment. Presumably, the response assessed at the 2nd MRI PET (before cycle 4 or induction chemotherapy) would be predictive of the overall response at the end of neoadjuvant treatment. Then, it would be possible to predict precociously the tumor response.

DETAILED DESCRIPTION:
The management of localized rectal cancer is done in two phases. The first phase, medical, combines a possible first chemotherapy, followed by a concomitant chemoradiotherapy. The second phase, 6 to 8 weeks later, consists of surgery of the rectum.

Magnetic resonance imaging (MRI) of the pelvis allows staging of the tumor and its possible lymph node extensions. MRI can also be used to assess tumor response after the first phase of treatment and before surgery. But MRI of the pelvis is partially imperfect.

PET-MRI is an examination that combines MRI with an injection of [18 F]fluorodeoxyglucose (18F-FDG). It is known to be more sensitive in assessing tumor stage and lymph node extensions compared to MRI and more sensitive in assessing tumor response before surgery.

The aim of this study is to determine predictive parameters for response to the first phase of treatment by accurately identifying the characteristics of tumors that have responded or not to treatment with chemotherapy and chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Histologically proven rectal cancer
* clinical tumor classification (cT) : cT3 - cT4 or all T / N+ / M0
* Tumor resectable or considered resectable after chemoradiotherapy
* Decision chemotherapy followed by neoadjuvant chemoradiotherapy decided at the organ Multidisciplinary Meeting
* Absence of distant metastases
* Adequate contraception for women of childbearing potential
* Adequate hematologic function
* Adequate liver function
* Free, signed and informed consent
* For women of childbearing potential : negative pregnancy test

Exclusion Criteria:

* Subject with Uncontrolled diabetes
* Contraindication to surgery
* Contraindication to MRI
* Contraindication to PET scan
* Contraindication to chemotherapy
* History of pelvic radiotherapy
* History of major co-morbidity that may prevent treatment and no active infection (HIV or chronic hepatitis B or C)
* Hypofractionated radiotherapy according to the Swedish protocol (25 Gy in 5 fractions)
* Colloid (mucinous) adenocarcinoma
* Presence of distant metastases
* Contraindication to 5-FluoroUracil (FU), oxaliplatin or irinotecan
* History of known Gilbert's disease
* Patient with known UGT1A1 genotype
* Known Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency
* Medical history of chronic diarrhea or inflammatory disease of the colon or rectum
* Medical history of angina or myocardial infarction.
* Active progressive infection or any other serious medical condition that could compromise the administration of the treatment
* Other concurrent cancer, or medical history of cancer other than treated in situ cervical carcinoma or basal cell carcinoma or squamous cell carcinoma
* Patient enrolled in another clinical trial testing an investigational agent
* Pregnant or breastfeeding woman
* Persons deprived of their freedom or under guardianship or incapable of giving consent
* Any psychological, familial, sociological or geographic condition that may interfere with the study protocol or follow-up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with histologically proven rectal cancer with an indication for induction chemotherapy followed by neoadjuvant chemoradiotherapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Description of the correlation between the PET-MRI changes after neo-adjuvant treatment and the histological response after surgery in terms of metabolic criteria. | At the surgery
  The purpose of this study is to determine predictive parameters for response to the first phase of treatment by accurately identifying the characteristics of tumors that have responded or not to chemotherapy and chemoradiotherapy.
  Metabolic criteria will be measured with the SUVmax values that will be determined on the 4 PET-MRI scans.
Description of the correlation between the PET-MRI changes after neo-adjuvant treatment and the histological response after surgery in terms of MRI criteria. | At the surgery
  MRI criteria will be measured with the Apparent Diffusion Coefficient (ADC) values that will be determined on the 4 PET-MRI scans.
Description of the correlation between the PET-MRI changes after neo-adjuvant treatment and the histological response after surgery in terms of anatomopathological criteria. | At the surgery
  Anatomopathological criteria will be measured with the histopathological response to treatment which will be defined according to the tumor regression grade (TRG)

SECONDARY OUTCOMES:
Comparison of the first PET-MRI staging with standard of care imaging, namely pelvic MRI in terms of tumor volumes | At the PET MRI pretherapy (= PET MRI 1)
  Record of tumor volumes on MRI PET 1
Comparison of the first PET-MRI staging with standard of care imaging, namely pelvic MRI in terms of SUVmax values | At the PET MRI pretherapy (= PET MRI 1)
  Record of SUVmax on MRI PET 1
Comparison of the first PET-MRI staging with standard of care imaging, namely pelvic MRI in terms of ADC values | At the PET MRI pretherapy (= PET MRI 1)
  Record of ADC on MRI PET 1
Description of the specific PET-MRI responses at mid-treatment of the neoadjuvant chemotherapy in terms of delta tumor volume | At the 2nd PET (PET2), up to 28 months
  Record of delta tumor volume, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses at mid-treatment of the neoadjuvant chemotherapy in terms of delta SUVmax values | At the 2nd PET (PET2), up to 28 months
  Record of delta SUVmax, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses at mid-treatment of the neoadjuvant chemotherapy in terms of delta ADC values | At the 2nd PET (PET2), up to 28 months
  Record of delta ADC, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses to neoadjuvant chemotherapy in terms of delta tumor volume | At the 3rd PET (PET3), up to 28 months
  Record of delta tumor volume, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses to neoadjuvant chemotherapy in terms of delta SUVmax values | At the 3rd PET (PET3), up to 28 months
  Record of delta SUVmax, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses to neoadjuvant chemotherapy in terms of delta ADC values | At the 3rd PET (PET3), up to 28 months
  Record of delta ADC, compared to baseline (PET MRI 1)
Description of the specific PET-MRI responses to neoadjuvant radiochemotherapy in terms of delta tumor volume | At the 4th PET (PET4), up to 28 months
  Record of delta tumor volume, compared to PET3
Description of the specific PET-MRI responses to neoadjuvant radiochemotherapy in terms of delta SUVmax values | At the 4th PET (PET4), up to 28 months
  Record of delta SUVmax, compared to PET3
Description of the specific PET-MRI responses to neoadjuvant radiochemotherapy in terms of delta ADC values | At the 4th PET (PET4), up to 28 months
  Record of delta ADC, compared to PET3
Propose standardized criteria to differentiate responders from non-responders | Data record throughout the study, up to 28 months
  Record of clinical and iconographic data predictive of good response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France